CLINICAL TRIAL: NCT01958697
Title: Age and Gender Corrected Body Mass Index: When Preoperative Weight Loss and Underweight Are Becomming Clinically Significant in Esophagectomy for Cancer.
Brief Title: Age and Gender Corrected Body Mass Index
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Johnny Moons, Datamanager Thoracic Surgery, University Hospital, Gasthuisberg
Other Study IDs: AG-BMI
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Esophageal Cancer
Keywords: Nutritional Disorders; Feeding Behavior
MeSH Terms: conditions — Esophageal Neoplasms; Nutrition Disorders; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AG-BMI < 10 pct: Patients who's peroperative BMI is less than the 10th centile
- AG-BMI >= 10th pct: Patients who's peroperative BMI equals or is greater than the 10th centile

SUMMARY:
Esophagectomy for cancer is often accompanied with severe preoperative weight loss. Body Mass Index (BMI) values are age-independent and the same for both sexes. From the perspective that these two parameters should actually be taken into account too, we developed a model to calculate "age-gender specific BMI-percentiles" (AG-BMI) and tested this model in relation to survival outcome after esophagectomy for cancer.

DETAILED DESCRIPTION:
Age-Gender specific BMI percentiles are more accurate compared to the current BMI classes in predicting Overall Survival (OS) after esophagectomy for cancer. Furthermore we believe in a more devastating impact on OS from underweight and not from overweight.

By preoperatively identifying risk patients for poorer OS, especially the non-tumoral deaths, this can be a tool to tailor postoperative nutritional strategies to counter further weight loss and bringing postoperative weight to normal ranges.

ELIGIBILITY:
Inclusion Criteria:

* any type of esophagectomy

Exclusion Criteria:

* Preoperative organ metastasis (cM+ or yM+)
* esophageal bypass surgery

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal cancer patients recieving an esophagectomy
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-10 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Overall 5 year survival | 5 years after esophagectomy
  Overall 5-year survival after esophagectomy for cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Univresity Hospital Leuven - dept. Thoracic Surgery, Leuven, Belgium